CLINICAL TRIAL: NCT06355414
Title: Psilocybin and Affective Function in Chronic Lower Back Pain Depression
Brief Title: Psilocybin in Chronic Low Back Pain and Depression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00385932; R33AT012317 (NIH)
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low-back Pain; Depression
Keywords: Psilocybin; Chronic Low-back Pain; Depression
MeSH Terms: conditions — Depression | interventions — Psilocybin; Methylphenidate

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, active control study comparing the effects of psilocybin (25mg fixed dose) and methylphenidate (40mg fixed dose)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial, and efforts will be made to mask the study drug (psilocybin) and the active control (methylphenidate) from participants, guides, and study staff. Participants will be debriefed about their randomly assigned drug condition after the completion of the final follow-up assessment, or after discontinuation/withdrawal, whichever comes first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): This arm will receive a single, absolute dose (25 mg) of psilocybin.
  Interventions: Drug: Psilocybin
- Methylphenidate (Active Comparator): This arm will receive a single, absolute dose (40 mg) of methylphenidate.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Psilocybin — Drug administration under supportive conditions
  Arms: Psilocybin
Drug: Methylphenidate — Drug administration under supportive conditions
  Arms: Methylphenidate

SUMMARY:
This study seeks to provide insight on psilocybin's effects on mechanisms of chronic pain among patients with co-morbid chronic low back pain and depression (CLBP+D).

Participants will receive either a single high-dose of psilocybin (25mg absolute dose) or methylphenidate (40mg absolute dose). Participants will be asked to complete assessments of pain, depressive symptoms, and more general questionnaires regarding the participants experiences during the experimental sessions and the associated enduring effects.

DETAILED DESCRIPTION:
This study will investigate the effects of a single experimental psilocybin (25 mg fixed dose) administration compared to a dose of methylphenidate (40 mg fixed dose). Assessments will be conducted during screening visits, before and after the drug session, at follow up visits up to 1-month after the drug session, as well as periodically throughout study participation via a multi-time-per-day survey application. Forty participants will complete all study visits including follow-up visits.

Primary objectives:

1. Investigate the feasibility, safety, and acceptability of psilocybin for CLBP+D
2. Investigate the effect of psilocybin on self-report of positive affect, negative affect, and pain catastrophizing
3. Investigate the effect of psilocybin on a behavioral task called positive affective pain inhibition

Secondary objectives:

1. Investigate the durability (1-month follow-up) effects of psilocybin on self-report of positive affect, negative affect, and pain catastrophizing
2. Investigate the effect of psilocybin on dynamic associations between affective measures, pain, and function on a moment-to-moment basis.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 80 years old
* Have given written informed consent
* Report low back pain as ongoing problem ≥ 3 months and any low back pain on at least half of the days over the past 6 months (consistent with NIH Consensus Recommendations for defining CLBP; other chronic pain problems can be present, but CLBP must be reported as primary)
* Report at least moderate depression symptoms Grid-Hamilton Depression Rating Scale (GRID-HAMD) ≥ 17
* Fluent in English
* At least high school level of education
* Agree to abstain from any psychoactive drugs on the day prior to and the day of the drug administration session
* Women who are of childbearing potential and sexually active who are not practicing an effective means of birth control must agree to practice an effective means of birth control throughout the duration of the study
* Be judged by study team clinicians to be at low risk for suicidality
* Concurrent psychotherapy or pharmacotherapy with selective serotonin reuptake inhibitors (SSRIs), serotonin and norephinephrine reuptake inhibitors (SNRIs), and/or bupropion (< 300 mg bupropion) is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study.
* Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study
* Be otherwise medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests; CBC, comprehensive metabolic panel (CMP), urine beta-human chorionic gonadotropin (HCG), urine toxicology screen.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree not to take any as needed (PRN) medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Have limited lifetime use of hallucinogens (the following criteria are preferred: no use in the past 5 years; total hallucinogen use less than 10 times)

Exclusion Criteria:

* Lifetime history of serious psychiatric (other than depression) or neurological disorders, including bipolar disorder, psychosis, or seizure disorder
* History (past 2 years) of severe substance use disorder or current (past six months) substance use disorder of moderate severity
* Clinically significant suicidal ideation (e.g. with strong intent or means) within past 6 months or history (past 5 years) of suicide attempt
* Medical condition incompatible with psilocybin administration (e.g., cardiovascular)
* On unstable/changing dose of opioid, benzodiazepine or other psychoactive or pain medication within 4 weeks prior to enrollment and/or unable to abstain from medication on drug administration day
* Current use/positive toxicology for illicit drugs or positive breath alcohol test at screening and prior to each drug administration session.
* Clinically significant transaminitis- aspertate aminotransferase (AST) or alanine aminotransferase (ALT) greater than two times normal value).
* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing;
* Women who are of childbearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged corrected QT interval (QTc) interval (i.e., QTc > 450 msec), heart valve, or transient ischemic attack (TIA) in the past year.
* History of seizures and/or epilepsy with history of seizures.
* Type 1 diabetes.
* BMI < 18
* Medical conditions contraindicated for methylphenidate administration:

  1. Concomitant use of Monoamine oxidase inhibitors (MAOIs), or use within 14 days of MAOI discontinuation
  2. Family history or diagnosis of Tourette's syndrome
  3. Known Fructose intolerance, glucose-galactose malabsorption, or sucrase-isomaltose insufficiency
  4. Glaucoma
  5. Known hypersensitivity to methylphenidate
  6. Marked agitation, anxiety, and tension
  7. Motor tics
* Currently taking on a regular (e.g., daily) basis any antidepressant medications other than SSRIs, SNRIs, or bupropion, or any other medications that have a primary centrally-acting serotonergic effect, including MAOIs. Bupropion dosage must be < 300 mg in order to be included. For individuals who have intermittent or PRN use of such medications and/or who taper off such medications after regular use, psilocybin sessions will not be conducted until at least 14 days or 5 half-lives (whichever is greater) of the agent have elapsed after the last dose.
* Nicotine dependence that would be incompatible with an individual to be nicotine free for 8-10 hours on a psilocybin session day
* Have a first degree relative with schizophrenia or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I disorder

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in positive affect as assessed by discrete positive affect items and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA Post-drug Session (1-day through 1-week after drug session) relative to Baseline (beginning the day after baseline visit is complete)
  Discrete positive affect items: joy, love, hope, contentment. Positive affect will be assessed by asking participants to rate the intensity of four discrete positive emotions (joy, love, hope, contentment) on a 5-point Likert scale from 1-5 ("Very slightly or not at all" to "Extremely") and averaging those discrete items. Positive Affect scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Higher Positive Affect scores represent higher levels of positive affect.
  A separate set of linear mixed-effects models (LMERs) will be utilized for each primary endpoint (aggregated averages of momentary positive affect), with a primary LMER estimating the difference between Baseline and Week 1. The Time x Group interaction will be the primary focus, and we aim to evaluate 1) the extent to which the primary endpoint differs between Baseline and Week 1, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in negative affect as assessed by discrete negative affect items and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA Post-drug Session (1-day through 1-week after drug session) relative to Baseline (beginning the day after baseline visit is complete)
  Discrete negative emotion items: depressed, angry, frustrated, and worried. Negative affect will be assessed by asking participants to rate the intensity of four discrete negative emotions (depressed, angry, frustrated, and worried) on a 5-point Likert scale from 1-5 ("Very slightly or not at all" to "Extremely") and averaging those discrete items. Negative Affect scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Lower Negative Affect scores represent lower levels of negative affect.
  A separate set of LMERs will be utilized for each primary endpoint (aggregated averages of momentary negative affect), with a primary LMER estimating the difference between Baseline and Week 1. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the primary endpoint differs between Baseline and Week 1, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in Pain Catastrophizing as assessed by the Pain Catastrophizing Scale and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA Post-drug Session (1-day through 1-week after drug session) relative to Baseline (beginning the day after baseline visit is complete)
  Pain catastrophizing will be assessed with three items taken from the Pain Catastrophizing Scale that have been specifically validated for use in Ecological Momentary Assessment (EMA) studies of patients with chronic pain. Items will be administered via EMA and scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Each item is on a 5-point Likert scale (ranging from 0, "Not at all", to 4, "All the time"). Higher scores on each of these items indicates increased pain catastrophizing.
  A separate set of LMERs will be utilized for each primary endpoint (aggregated averages of momentary pain catastrophizing), with a primary LMER estimating the difference between Baseline and Week 1. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the primary endpoint differs between Baseline and Week 1, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in Positive Affective Pain Inhibition (Quantitative Sensory Testing) | Baseline, 1-week follow-up
  Positive Affective Pain Inhibition will be assessed using quantitative sensory testing at baseline, 1-week post-drug-administration, and 1-month post-drug-administration. Positive affective pain inhibition is measured as the difference in pain ratings to noxious stimuli administered during the presentation of positive/rewarding stimuli relative to neutral or negative stimuli.
  A separate set of LMERs will be utilized for each primary endpoint (index of Positive Affective Pain Inhibition), with a primary LMER estimating the difference between Baseline and Week 1. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the primary endpoint differs between Baseline and Week 1, and 2) the extent to which that difference varies between the Psilocybin and Control groups.

SECONDARY OUTCOMES:
Changes in positive affect as assessed by discrete positive affect items and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA 1-month Post-drug (7 days leading up to 1-month follow-up) relative to Baseline (beginning the day after baseline visit is complete)
  Discrete positive affect items: joy, love, hope, contentment. Positive affect will be assessed by asking participants to rate the intensity of four discrete positive emotions (joy, love, hope, contentment) on a 5-point Likert scale from 1-5 ("Very slightly or not at all" to "Extremely") and averaging discrete items. Positive Affect scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Higher Positive Affect scores represent higher levels of positive affect.
  A separate set of LMERs will be utilized for each endpoint (aggregated averages of momentary positive affect), with a secondary LMER estimating the difference between Baseline and 1-Month. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the secondary endpoint differs between Baseline and 1-Month, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in negative affect as assessed by discrete negative affect items and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA 1-month Post-drug (7 days leading up to 1-month follow-up) relative to Baseline (beginning the day after baseline visit is complete)
  Discrete negative emotion items: depressed, angry, frustrated, and worried. Negative affect will be assessed by asking participants to rate the intensity of four discrete negative emotions (depressed, angry, frustrated, and worried) on a 5-point Likert scale from 1-5 ("Very slightly or not at all" to "Extremely") and averaging discrete items. Negative Affect scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Lower Negative Affect scores represent lower levels of negative affect.
  A separate set of LMERs will be utilized for each endpoint (aggregated averages of momentary negative affect), with a secondary LMER estimating the difference between Baseline and 1-Month. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the secondary endpoint differs between Baseline and 1-Month, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in Pain Catastrophizing as assessed by the Pain Catastrophizing Scale and averaged over 7-day periods of Ecological Momentary Assessment (EMA) | 7-day period of EMA 1-month Post-drug (7 days leading up to 1-month follow-up) relative to Baseline (beginning the day after baseline visit is complete)
  Pain catastrophizing will be assessed with three items taken from the Pain Catastrophizing Scale that have been specifically validated for use in Ecological Momentary Assessment (EMA) studies of patients with chronic pain. Items will be administered via EMA and scores will be aggregated over 7-day EMA periods at baseline, post-session, and 1-month follow-up. Each item is on a 5-point Likert scale (ranging from 0, "Not at all", to 4, "All the time"). Higher scores on each of these items indicates increased pain catastrophizing.
  A separate set of LMERs will be utilized for each endpoint (aggregated averages of momentary pain catastrophizing), with a secondary LMER estimating the difference between Baseline and 1-Month. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the secondary endpoint differs between Baseline and 1-Month, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Changes in Positive Affective Pain Inhibition (Quantitative Sensory Testing) | Baseline, 1-Month follow-up
  Positive Affective Pain Inhibition will be assessed using quantitative sensory testing at baseline, 1-week post-drug-administration, and 1-month post-drug-administration. Positive affective pain inhibition is measured as the difference in pain ratings to noxious stimuli administered during the presentation of positive/rewarding stimuli relative to neutral or negative stimuli.
  A separate set of LMERs will be utilized for each endpoint (index of Positive Affective Pain Inhibition), with a secondary LMER estimating the difference between Baseline and 1-Month. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the secondary endpoint differs between Baseline and 1-Month, and 2) the extent to which that difference varies between the Psilocybin and Control groups.

OTHER OUTCOMES:
Pain as assessed by discrete pain items assessed via EMA | 7-day periods of EMA at 1-week follow-up and 1-month follow-up, each relative to Baseline
  Discrete pain items include 'Rate your current level of pain' and 'Over the past hour: Rate the worst pain you experienced.' These items will be assessed multiple times daily during each EMA items. These items will be averaged over each EMA burst to determine pain levels over the course of trial participant.
  A separate set of LMERs will be utilized for each endpoint (aggregated averages of momentary pain ratings), with LMERs estimating the differences between Baseline and 1-Week as well as 1-Month. The Time x Group interaction will be the primary focus of interest, and we aim to evaluate 1) the extent to which the endpoint differs between Baseline and 1-Week as well as 1-Month, and 2) the extent to which that difference varies between the Psilocybin and Control groups.
Dynamic association between affect and pain using micro-longitudinal EMA data of affective variables (positive, negative affect outcomes) and pain outcomes | 7-day periods of EMA at: Baseline (beginning the day after baseline visit is complete), Post-drug Session (beginning the day after drug session), and 1-month follow-up (the seven days leading up to the 1-month follow-up visit)
  Our secondary analytic strategy will focus on the dynamic association between affect and pain using the micro-longitudinal EMA data, in which the EMA data is organized hierarchically with Waves (Baseline, 1-week, 1-month) nested within People, Days nested within Waves, and Momentary Observations (up to four) nested within Days. For each EMA wave (Baseline, 1-week, and 1-month), we will utilize separate LMERs to evaluate the momentary (i) concurrent and (ii) lagged associations between affective variables and pain. In each LMER, person-mean centered day-level affective variables and Group (Psilocybin vs. Methylphenidate) will be included as fixed effects; day-level intercept and participant-level intercept will be included as random effects. Results from these LMERs will also allow us to evaluate the extent to which the momentary concurrent/lagged associations differ by group at each EMA wave.
Changes in mood as measured by a selection of discrete items derived from the Positive and Negative Affect Schedule- Expanded Form (PANAS-X). | 7-day periods of EMA at: Baseline (beginning the day after baseline visit is complete), Post-drug Session (beginning the day after drug session), and 1-month follow-up (the seven days leading up to the 1-month follow-up visit)
  The selected, discrete positive and negative affect items described in Primary Outcome 1 will be supplemented by a selection of discrete items derived from the Positive and Negative Affect Schedule- Expanded Form (PANAS-X) and measured via Ecological Momentary Assessment (EMA).
Changes in self-reported Pain Impact as measured by Pain intensity (P), interference with Enjoyment of life (E), and interference with General activity (G) Scale (PEG) | 7-day periods of EMA at: Baseline (beginning the day after baseline visit is complete), Post-drug Session (beginning the day after drug session), and 1-month follow-up (the seven days leading up to the 1-month follow-up visit)
  Pain impact will be assessed with the Pain average, interference with Enjoyment of life, and interference with General activity (PEG), which will be assessed with EMA over the course of three distinct 7-day periods at baseline, immediately following drug session, and leading up to 1-month follow-up to permit time-varying analyses of the associations of affective mechanisms with pain and function. The PEG is a three-item measure scored, with each item rated on a scale of 0-10. Higher scores indicate higher levels of pain intensity or higher levels of interference of interference with enjoyment/general activity, depending on the item. Overall, higher scores indicate higher levels of pain impact.
Changes in Pressure Pain Threshold (Quantitative Sensory Testing) | Baseline, 1-week follow-up, 1-month follow-up
  An electronic algometer with a 1cm2 hard rubber probe will be used to assess responses to noxious mechanical pressure, according to standard procedures. Pressure at the site is gradually increased at a steady rate and stopped when the subject indicates the stimulus is first perceived as painful and/or tolerance is reached.
Changes in Conditioned Pain Modulation (Quantitative Sensory Testing) | Baseline, 1-week follow-up, 1-month follow-up
  The thermal (primary outcome for determination of painful stimuli, as in Primary Outcome 3) and pressure (secondary outcome for pain testing, described in Outcome 16) stimuli may be presented together or in succession to assess conditioned pain modulation.
Chronic Pain Exacerbation as measured by the Graded Chronic Pain Scale- Revised (GCPS-R) | Baseline, 1-week follow-up, 1-month follow-up
  Chronic Pain Exacerbation will be assessed via the Graded Chronic Pain Scale- Revised (GCPS-R). This scale probes the frequency of pain and the degree to which it interferes with daily life and work activities. Responding that the pain interferes more frequently results in a higher a grade. The GCPS-R is graded from 0 (Chronic Pain Absent) to 3 (High-Impact Chronic Pain).
Changes in neuropathic pain features as assessed by the painDETECT questionnaire (PDQ) | Baseline, 1-week follow-up, 1-month follow-up
  Neuropathic pain features will be assessed with the painDETECT questionnaire (PDQ). The PDQ comprises 12 items. The resulting total score classifies pain into three groups: a score > 18 indicates that the presence of a predominant neuropathic pain component is likely, a score of 13 to 18 is considered uncertain, and a score < 13 indicates that a neuropathic pain component is not likely present.
Changes in CLBP-related disability as measured by the Oswestry Disability Index (ODI) | Baseline, 1-week follow-up, 1-month follow-up
  CLBP-related disability will be assessed with the Oswestry Disability Index (ODI). The ODI is a self-administered questionnaire divided into ten sections/items designed to assess limitations of various activities of daily living. Patients are asked to select which statement they agree with most on each item/section of the index, and each section is scored on a 0-5 scale, 5 representing the greatest disability. Summed scores range from 0-50, with 0 representing "no disability" and 50 representing "completely disabled".
Change in Emotion Regulation as assessed by the Difficulties in Emotion Regulation Scale (DERS) | Baseline, 1-week follow-up, 1-month follow-up
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale (DERS). This is self-report scale that asks respondents how they relate to their emotions. Items are rated on a scale of 1 ("almost never") to 5 ("almost always"). Higher scores indicate more difficulty in emotion regulation.
Pain intensity and related dimensions of health (i.e., sleep) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS-29 v2.0). | Baseline, 1-week follow-up, 1-month follow-up
  The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. Higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function).
Psychological Inflexibility in Pain as measured by the Psychological Inflexibility in Pain Scale (PIPS) | Baseline, 1-week follow-up, 1-month follow-up
  Psychological Inflexibility in Pain. The PIPS is a 12-item questionnaire that aims at measuring psychological inflexibility with two subscales, Avoidance of Pain (Avoidance) and Cognitive Fusion with Pain (Fusion). The PIPS consists of 12 items rated on a 7-point scale from 1 (never true) to 7 (always true). Higher scores indicate greater levels of psychological inflexibility.
Personal values and the degree of success in following those values as measured by the Chronic Pain Values Inventory (CPVI). | Baseline, 1-week follow-up, 1-month follow-up
  The 12-item CPVI is a brief inventory that can be used to determine which values are important to an individual and to assess the degree of success they are having in following their values. The valued domains included in the inventory are family, intimate relations, friends, work, health, and growth or learning. Participants will be asked to rate each item on a scale from 0 (not at all important / successful) to 5 (extremely important / successful). Two primary scores are obtained when scoring the CPVI. The first is a mean success rating, taken as the average of the 6 success ratings. The second score is a mean discrepancy rating, taken as the mean of the differences between importance and success.
Dispositional tendencies to feel positive emotions towards others in daily life as measured by the Dispositional Positive Emotion Scale (DPES) | Baseline, 1-week follow-up, 1-month follow-up
  Dispositional Positive Emotion Scale (DPES) consists of seven subscales (joy, contentment, pride, love, compassion, amusement and awe) that measure dispositional tendencies to feel positive emotions towards others in daily life. There are 38 items in total, each on a 7-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (7). Items are averaged, yielding a total score ranging from 1 to 7. Higher scores indicate greater levels of positive emotion.
Mindfulness as measured by the Five Facet Mindfulness Questionnaire (FFMQ-15) | Baseline, 1-week follow-up, 1-month follow-up
  Five Facet Mindfulness Questionnaire (FFMQ-15) measures mindfulness across five subscales and is used in clinical practice to assess the effect of mindfulness on psychological health. The five subscales are: observing, describing, acting with awareness, non-judgment, and non-reactivity. Results consist of a total average score and five subscale scores. Average scores are calculated by summing the responses and dividing by the number of items, and indicate the average level of agreement with the each subscale (1 = rarely true, 5 = always true). Higher scores are indicative of someone who is more mindful in their everyday life.
Subjective experiences: Awe Experience Scale (AWE-S) | post drug administration up to 8 hours, 1-week follow-up, 1-month follow-up
  The subjective experience of the drug will also be assessed with the Awe Experience Scale. Items are scored on a 7-point Likert scale, and a higher score indicates individuals experience the emotion of awe more often.
Subjective experiences: Mystical Experience Questionnaire (MEQ30) | post drug administration up to 8 hours, 1-week follow-up, 1-month follow-up
  The subjective experience of the drug will be assessed with the Mystical Experience Questionnaire. The MEQ30 is a 30-item questionnaire assessing mystical-type experiences (typically following psilocybin or other psychedelic drug sessions). Higher scores on this measure reflect higher incidence of mystical experiences.
Subjective experiences: Challenging Experience Questionnaire (CEQ) | post drug administration up to 8 hours, 1-week follow-up, 1-month follow-up
  The subjective experience of the drug will also be assessed with the Challenging Experience Questionnaire (CEQ), a 26-item measure assessing seven dimensions of psychedelic-occasioned challenging experiences: grief, fear, death, insanity, isolation, physical distress, and paranoia. Response are on 6-point scale from 0, "None/not at all" to 5 "Extreme (more than ever before in my life)", indicating the degree to which the individual experienced each of a series of subjective effects during their drug session. Each item is divided by the maximum possible score; subscale scores are obtained by totaling all transformed items under that subscale to obtain each subscale score; total score is obtained by summing all transformed items on the questionnaire. Higher scores on both subscale and total scores indicate more challenging experiences.
Subjective experiences: Altered States of Consciousness Questionnaire (5D-ASC) | post drug administration up to 8 hours, 1-week follow-up, 1-month follow-up
  The subjective experience of the drug will also be assessed with the 5D-ASC, a 94-item self-report scale that assesses the participants' alterations from normal waking consciousness. Participants are asked to rate each item on a scale of "No, not more than usually" to "Yes, much more than usually," and higher scores reflect greater alterations from normal waking consciousness.
Subjective experiences: Psychological Insight Questionnaire (PIQ) | post drug administration up to 8 hours, 1-week follow-up, 1-month follow-up
  The subjective experience of the drug will also be assessed with the Psychological Insight Questionnaire (PIQ). The PIQ consists of 23 items with two subscales: (a) Avoidance and Maladaptive Patterns Insights and (b) Goals and Adaptive Patterns Insights. Responses are on a scale from 0, "No; not at all" to 5 "Extremely (more than ever before in my life)." Subscale scores and total scores are determined by computing the mean of all items under the individual subscales (PIQ subscale scores) or all items on the questionnaire (total PIQ score). Higher sub scale and total scores reflect greater psychological insight.
Changes in basic beliefs about the world as measured by the Primals Inventory (PI-6) | Baseline, 1-week follow-up, 1-month follow-up
  Primals Inventory (PI-6): A six-item scale that probes basic beliefs about the world. Items are scored on a six-point Likert scale, from 0 ('Strongly Disagree') to 5 ('Strongly Agree). Higher scores indicates greater alignment with the primal being measured.

CONTACTS AND LOCATIONS:
Overall Officials: David B Yaden, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak HW, Schneider S. Individual differences in momentary pain-affect coupling and their associations with mental health in patients with chronic pain. J Psychosom Res. 2020 Nov;138:110227. doi: 10.1016/j.jpsychores.2020.110227. Epub 2020 Aug 28. PMID 32919151
- [Background] Roy M, Peretz I, Rainville P. Emotional valence contributes to music-induced analgesia. Pain. 2008 Jan;134(1-2):140-7. doi: 10.1016/j.pain.2007.04.003. Epub 2007 May 25. PMID 17532141
- [Background] Sullivan MJ, Bishop SR, & Pivik J (1995). The pain catastrophizing scale: development and validation. Psychol Assess, 7(4): 524.
- [Background] Vanderlind WM, Everaert J, Joormann J. Positive emotion in daily life: Emotion regulation and depression. Emotion. 2022 Oct;22(7):1614-1624. doi: 10.1037/emo0000944. Epub 2021 Mar 4. PMID 33661667
- [Background] Yaden, D. B., Kaufman, S. B., Hyde, E., Chirico, A., Gaggioli, A., Zhang, J. W., & Keltner, D. (2019). The development of the Awe Experience Scale (AWE-S): A multifactorial measure for a complex emotion. The Journal of Positive Psychology, 14(4): 474-488.
- [Background] Kroenke K, Wu J, Bair MJ, Krebs EE, Damush TM, Tu W. Reciprocal relationship between pain and depression: a 12-month longitudinal analysis in primary care. J Pain. 2011 Sep;12(9):964-73. doi: 10.1016/j.jpain.2011.03.003. Epub 2011 Jun 16. PMID 21680251
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Griffiths RR, Richards WA, McCann U, Jesse R. Psilocybin can occasion mystical-type experiences having substantial and sustained personal meaning and spiritual significance. Psychopharmacology (Berl). 2006 Aug;187(3):268-83; discussion 284-92. doi: 10.1007/s00213-006-0457-5. Epub 2006 Jul 7. PMID 16826400
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology & Behavioral Assessment, 26(1): 41
- [Background] George SZ, Calley D, Valencia C, Beneciuk JM. Clinical Investigation of Pain-related Fear and Pain Catastrophizing for Patients With Low Back Pain. Clin J Pain. 2011 Feb;27(2):108-15. doi: 10.1097/AJP.0b013e3181f21414. PMID 20842009
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Flink IL, Boersma K, Linton SJ. Pain catastrophizing as repetitive negative thinking: a development of the conceptualization. Cogn Behav Ther. 2013;42(3):215-23. doi: 10.1080/16506073.2013.769621. PMID 23978106
- [Background] Finan PH, Garland EL. The role of positive affect in pain and its treatment. Clin J Pain. 2015 Feb;31(2):177-87. doi: 10.1097/AJP.0000000000000092. PMID 24751543
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Dittrich A. The standardized psychometric assessment of altered states of consciousness (ASCs) in humans. Pharmacopsychiatry. 1998 Jul;31 Suppl 2:80-4. doi: 10.1055/s-2007-979351. PMID 9754838
- [Background] Davis AK, Barrett FS, So S, Gukasyan N, Swift TC, Griffiths RR. Development of the Psychological Insight Questionnaire among a sample of people who have consumed psilocybin or LSD. J Psychopharmacol. 2021 Apr;35(4):437-446. doi: 10.1177/0269881120967878. Epub 2021 Jan 9. PMID 33427007
- [Background] Barrett FS, Johnson MW, Griffiths RR. Validation of the revised Mystical Experience Questionnaire in experimental sessions with psilocybin. J Psychopharmacol. 2015 Nov;29(11):1182-90. doi: 10.1177/0269881115609019. Epub 2015 Oct 6. PMID 26442957
- [Background] Barrett FS, Bradstreet MP, Leoutsakos JS, Johnson MW, Griffiths RR. The Challenging Experience Questionnaire: Characterization of challenging experiences with psilocybin mushrooms. J Psychopharmacol. 2016 Dec;30(12):1279-1295. doi: 10.1177/0269881116678781. Epub 2016 Nov 17. PMID 27856683
- [Background] McCracken LM, Yang SY. The role of values in a contextual cognitive-behavioral approach to chronic pain. Pain. 2006 Jul;123(1-2):137-45. doi: 10.1016/j.pain.2006.02.021. Epub 2006 Mar 29. PMID 16564627
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Clifton JDW, Yaden DB. Brief measures of the four highest-order primal world beliefs. Psychol Assess. 2021 Dec;33(12):1267-1273. doi: 10.1037/pas0001055. Epub 2021 Jul 1. PMID 34197163
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Nakonezny PA, Carmody TJ, Morris DW, Kurian BT, Trivedi MH. Psychometric evaluation of the Snaith-Hamilton pleasure scale in adult outpatients with major depressive disorder. Int Clin Psychopharmacol. 2010 Nov;25(6):328-33. doi: 10.1097/YIC.0b013e32833eb5ee. PMID 20805756
- [Background] Shiota, M. N., Keltner, D., & John, O. P. (2006). Positive emotion dispositions differentially associated with Big Five personality and attachment style. The Journal of Positive Psychology, 1(2), 61-71. DOI: 10.1080/17439760500510833
- [Background] Von Korff M, DeBar LL, Krebs EE, Kerns RD, Deyo RA, Keefe FJ. Graded chronic pain scale revised: mild, bothersome, and high-impact chronic pain. Pain. 2020 Mar;161(3):651-661. doi: 10.1097/j.pain.0000000000001758. PMID 31764390
- [Background] Wicksell RK, Lekander M, Sorjonen K, Olsson GL. The Psychological Inflexibility in Pain Scale (PIPS)--statistical properties and model fit of an instrument to assess change processes in pain related disability. Eur J Pain. 2010 Aug;14(7):771.e1-14. doi: 10.1016/j.ejpain.2009.11.015. Epub 2010 Jan 27. PMID 20106685
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039